CLINICAL TRIAL: NCT07327762
Title: COMPARISON OF TWO DIFFERENT SUTURE KNOT TECHNIQUES ON POST-OPERATIVE TRISMUS AND SWELLING AFTER IMPACTED THIRD MOLAR SURGERY
Acronym: Impacted molar
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Watim Medical & Dental College (Other)
Responsible Party: Principal Investigator, Shania Haq, Principal Investigator, Watim Medical & Dental College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WMDCR/ERB/2023/50
Record Dates: First submitted 2025-11-18; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Trismus; Swelling
MeSH Terms: conditions — Trismus

STUDY DESIGN:
Intervention Model Description: By undertaking a comparative analysis of two distinct suture knot techniques, this study seeks to address this knowledge gap and provide evidence-based insights into the optimal approach for wound closure in impacted third molar surgery. Understanding the differential effects of suture techniques on postoperative trismus and swelling is essential for informing clinical decision-making, guiding surgical practices, and ultimately enhancing patient care. Postoperative complications are common after this surgery and can be attributed to various factors.
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- locking suture (Experimental): effect of locking suture on trismus and swelling
  Interventions: Procedure: locking and non locking suture techniques; Procedure: non locking suture technique
- non locking suture (Experimental): effect of non locking suture on trismus and swelling
  Interventions: Procedure: locking and non locking suture techniques; Procedure: non locking suture technique

INTERVENTIONS:
Procedure: locking and non locking suture techniques — The participating patients will be randomly assigned into two groups, i.e. receiving locked (L) or unlocked (UL) sutures, using a lottery method. Equal patients will be assigned in both groups. In group L (Locked suturing), the flap will be repositioned and sutured with the locked technique (straight-reverse-straight) hermetically using 3-0 black silk. In group UL (Unlocked suturing), the flap will be repositioned and sutured with the unlocked technique (three straight knots) loosely using 3-0 black silk.
  Demographic details (including name, age, gender, contact) will be obtained and recorded on specific data collection forms.
  On the day of surgery before the surgery commences, measurements will be taken for trismus and swelling which will be entered on the data collection form.
  Trismus will be evaluated by measuring the distance between the mesio-incisal corners of the upper and lower right central incisors at maximum mouth opening in mm, using Castroviejo instrument.
  The facial swel
Procedure: non locking suture technique — The participating patients will be randomly assigned into two groups, i.e. receiving locked (L) or unlocked (UL) sutures, using a lottery method. Equal patients will be assigned in both groups. In group L (Locked suturing), the flap will be repositioned and sutured with the locked technique (straight-reverse-straight) hermetically using 3-0 black silk. In group UL (Unlocked suturing), the flap will be repositioned and sutured with the unlocked technique (three straight knots) loosely using 3-0 black silk. Demographic details (including name, age, gender, contact) will be obtained and recorded on specific data collection forms. On the day of surgery before the surgery commences, measurements will be taken for trismus and swelling which will be entered on the data collection form. Trismus will be evaluated by measuring the distance between the mesio-incisal corners of the upper and lower right central incisors at maximum mouth opening in mm, using Castroviejo instrument.

SUMMARY:
To compare the two different suture knot techniques, locked and unlocked, in terms of mean on postoperative trismus and swelling after impacted mandibular third molar surgery.

DETAILED DESCRIPTION:
The rationale behind conducting a comparative analysis of two different suture knot techniques on postoperative trismus and swelling following impacted third molar surgery stems from the imperative need to optimize patient outcomes and improve surgical practices. Impacted third molar surgery, while a routine procedure in oral and maxillofacial surgery, often presents challenges in managing postoperative complications, particularly trismus and swelling, which can significantly impact patients' comfort, recovery, and overall satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* • Healthy individuals

  * Gender: male and female
  * Age: 18-45 years
  * Mandibular third molar impaction all positions
  * Mandibular third molar impaction all classes

Exclusion Criteria:

* • Patients with ASA status III and above

  * Patients requiring multiple extractions in same appointment
  * Patients allergic to Lignocaine
  * Patients in whom adrenaline is contraindicated
  * Medically compromised individual such as those with poorly controlled diabetes, hypertension and pregnancy, etc.

Max Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
effect of locking and non locking suture technique on trismus | 3 days and 7 days post operatively
  Trismus will be evaluated by measuring the distance between the mesio-incisal corners of the upper and lower right central incisors at maximum mouth opening in mm, using Castroviejo instrument.
Effect of locking and unlocking sutures on facial swelling | Post operative day three and day seven
  The facial swelling in cm will be determined by measuring the distance from the corner of the mouth to the attachment of the earlobe following the bulge of the cheek and the distance from the outer canthus of the eye to the angle of the mandible using a plastic measuring tape.

CONTACTS AND LOCATIONS:
Locations (1):
- Watim Medical and Dental College, Rawalpindi, Pakistan, Pakistan